CLINICAL TRIAL: NCT01688154
Title: Ability of Grape Seed Proanthocyanidins to Reduce Postprandial Triglycerides in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: University Rovira i Virgili (Other); Hospital Universitari Sant Joan de Reus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 306724
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Triglyceride Metabolism; Cardiovascular Function
MeSH Terms: interventions — Grape Seed Proanthocyanidins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Product 1 (Active Comparator): 35 mg/Kg of grape seed proanthocyanidins extract (2 capsules)
  Interventions: Dietary Supplement: 35 mg/Kg of grape seed proanthocyanidins extract (2 capsules)
- Control product (Placebo Comparator): 2 empty capsules
  Interventions: Other: 2 empty capsules

INTERVENTIONS:
Dietary Supplement: 35 mg/Kg of grape seed proanthocyanidins extract (2 capsules)
  Arms: Product 1
Other: 2 empty capsules
  Arms: Control product

SUMMARY:
Grape seed proanthocyanidins have been reported to possess a hypotriglyceridemic effect after an acute or chronic consumption in rodents. In this study, we aimed to investigate the effects of an acute consumption of proanthocyanidins before a breakfast meal in humans. Moreover, the mechanisms implicated in the reduction of plasma triglycerides levels by grape seed proanthocyanidins in humans should be elucidated as well as its activity on vascular function.

DETAILED DESCRIPTION:
The intervention will consist in the administration of 2 capsules containing the grape seed proanthocyanidins extract or 2 empty capsules (placebo) just before breakfast, which will consist of 100g of white bread, 75g of salami, 50g of fatty cheese, 125g of yogurt (10% fat), 25ml of olive oil and water ad libitum. The nutritional composition of this meal is as follows: 1.200 Kcal of energy content, 15% of energy from proteins, 22% from carbohydrates and 63% from fat (35% saturated fat), and 120mg of cholesterol. Blood samples will be taken at point 0.5,1,2,3 and 6 hours after breakfast. Moreover, urine samples will be collected at time 0 and 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 20 and 40
* Signing the informed consent

Exclusion Criteria:

* Body mass index (BMI) lower than 18.5 or greater than 27 Kg/m2
* Smokers
* Regular medication
* Consumption of medication during the last week
* Following a weight-loss diet
* Vegetarians
* Abnormal glucose levels
* Diabetes
* Cardiovascular disease
* Gastrointestinal disease
* Anemia
* Nuts allergy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve of plasma triglycerides concentration | 0-180 minutes

SECONDARY OUTCOMES:
Blood pressure | 0-0.5-1-2-3-6 hours
Endothelial function (assessed by ischemic reactive hyperemia) | 0-0.5-1-2-3-6 hours
Blood lipid levels, markers of inflammation and oxidation | 0-0.5-1-2-3-6 hours
Plasma levels of procyanidins metabolites | 0-0.5-1-2-3-6 hours
Markers of cholesterol metabolism in PBMCs (mRNA and protein). | 0-0.5-1-2-3-6 hours
Membrane lipid composition of erythrocytes and oxidation markers. | 0-0.5-1-2-3-6 hours
Non-targeted metabolomics and 8-epi-prostaglandin-F2α levels (in urine) | 0-6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, PhD, Principal Investigator — University Rovira i Virgili; Maria Cinta Bladé, PhD, Principal Investigator — University Rovira i Virgili
Locations (2):
- Spain (2):
  - CTNS, Reus, Tarragona
  - Technological Center of Nutrition and Health (CTNS), Reus, Tarragona